CLINICAL TRIAL: NCT01494961
Title: The Public Health Impact of Couple-oriented Prenatal HIV Counseling in Low and Medium HIV Prevalence Countries
Brief Title: Couple-oriented Prenatal HIV Counseling in Low and Medium HIV Prevalence Countries
Acronym: Prenahtest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12127 Prenahtest
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Partner HIV Testing; Couple HIV Counseling; Couple Communication; HIV Incidence
Keywords: Partner HIV testing; Couple HIV counseling; Couple communication on sexual and reproductive health; HIV incidence; Incidence of pregnancies; Disclosure; Condom use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couple-oriented post-test HIV counseling (Experimental): Women received couple-oriented post-test HIV counseling
  Interventions: Behavioral: Couple-oriented post-test HIV counseling
- Standard post-test HIV counseling (No Intervention): Women received post-test HIV counseling as per standard site protocol

INTERVENTIONS:
Behavioral: Couple-oriented post-test HIV counseling — COC is an individual behavioural intervention, strengthening standard post-test HIV counselling delivered to pregnant women after prenatal HIV testing. COC was based on the assumption that developing women's communication skills and self-efficacy during HIV counselling would enable them to discuss HIV and sexual issues with their partners, and yield tangible effects on partner HIV testing. The structure of the COC intervention was adapted from a WHO PMTCT counselling manual and was described in a COC manual, which was used to train the COC counsellors and could also be used during the counselling session. Tested during the pilot phase of the trial, COC was shown to be feasible and acceptable in the four study sites.
  Arms: Couple-oriented post-test HIV counseling

SUMMARY:
ANRS 12127 Prenahtest is an intervention trial conducted in four countries (Cameroon, Dominican Republic, Georgia and India), where pregnant women are randomized during prenatal care to receive either standard post-test HIV counseling, or an innovative intervention called couple-oriented post-test HIV counseling (COC).

The aim of the COC intervention is to empower women to communicate with her male partner about HIV, and HIV testing in particular, and encourage him to return for HIV testing and/or couple HIV counseling (where both couple members are counseled together).

Prenahtest is the first randomised trial testing a prenatal intervention to increase partner HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* Attending her first ANC visit for the current pregnancy in the study centre
* Accepting to participate in the study and being able to give informed consent ii
* Currently having a partner (the man who the woman considers as her regular partner on the day of inclusion, even if this person is not the baby's father) iii
* Accepting follow-up (including home visits if necessary) by the project staff until 15 months after delivery

Exclusion Criteria:

* Having been tested for HIV during her current pregnancy
* Having a male partner who was tested for HIV during her gestational period v
* Having a partner who works out of the predefined study area or is absent for more then 6 months
* Being unwilling/unable to provide address/contact information
* Having an intoxication and/or mental impairment at the moment of recruitment

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1943 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Partner HIV testing | 6 months postpartum
  Proportion of male partners tested for HIV during the study follow-up period (from post-test HIV counseling to the last follow-up visit at 6 months postpartum) among the pregnant women enrolled in the trial

SECONDARY OUTCOMES:
Couple HIV counseling | 6 months postpartum
  Proportion of women receiving couple HIV counseling uring the study follow-up period (from post-test HIV counseling to the last follow-up visit at 6 months postpartum) among the pregnant women enrolled in the trial
HIV incidence | 6 months postpartum
  Proportion of women tested HIV-positive during the study follow-up period (from post-test HIV counseling to the last follow-up visit at 6 months postpartum) among the pregnant women tested HIV-negative at enrolment
Couple communication of sexual and reproductive health | 6 months postpartum
  Proportion of women reporting having discussed sexual and reproductive health issues (family planning, HIV, condom) during the study follow-up period (from post-test HIV counseling to the last follow-up visit at 6 months postpartum) among the pregnant women enrolled in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Francois Dabis, MD - PhD, Principal Investigator — INSERM U897, Institut de Santé Publique Epidémiologie Développement; Patrice T Tchendjou, MD - MPH, Principal Investigator — Centre Pasteur du Cameroon
Locations (4):
- Centre Mère - Enfant Chantal Biya, Yaoundé, Cameroon
- Hospital Materno-Infantil "San Lorenzo" de los Mina, Santo Domingo, Dominican Republic
- Maternity Hospital N°5, Tbilisi, Georgia
- Sane Guruji Hospital, Pune, India

REFERENCES:
- [Result] Orne-Gliemann J, Tchendjou PT, Miric M, Gadgil M, Butsashvili M, Eboko F, Perez-Then E, Darak S, Kulkarni S, Kamkamidze G, Balestre E, du Lou AD, Dabis F. Couple-oriented prenatal HIV counseling for HIV primary prevention: an acceptability study. BMC Public Health. 2010 Apr 19;10:197. doi: 10.1186/1471-2458-10-197. PMID 20403152
- [Result] Tchendjou PT, Koki PN, Eboko F, Malateste K, Essounga AN, Amassana D, Mossus T, Tejiokem M, Boisier P, Orne-Gliemann J. Factors associated with history of HIV testing among pregnant women and their partners in Cameroon: baseline data from a Behavioral Intervention Trial (ANRS 12127 Prenahtest). J Acquir Immune Defic Syndr. 2011 Jul 1;57 Suppl 1:S9-15. doi: 10.1097/QAI.0b013e31821ec6e2. PMID 21857289
- [Derived] Kengne-Nde C, Tejiokem MC, Orne-Gliemann J, Melingui B, Koki Ndombo P, Essounga NA, Bissek AC, Cauchemez S, Tchendjou PT. Couple oriented counselling improves male partner involvement in sexual and reproductive health of a couple: Evidence from the ANRS PRENAHTEST randomized trial. PLoS One. 2021 Jul 30;16(7):e0255330. doi: 10.1371/journal.pone.0255330. eCollection 2021. PMID 34329355
- [Derived] Tiendrebeogo T, Plazy M, Darak S, Miric M, Perez-Then E, Butsashvili M, Tchendjou P, Dabis F, Orne-Gliemann J. Couples HIV counselling and couple relationships in India, Georgia and the Dominican Republic. BMC Public Health. 2017 Nov 25;17(1):901. doi: 10.1186/s12889-017-4901-8. PMID 29178852
- [Derived] Orne-Gliemann J, Balestre E, Tchendjou P, Miric M, Darak S, Butsashvili M, Perez-Then E, Eboko F, Plazy M, Kulkarni S, Desgrees du Lou A, Dabis F; Prenahtest ANRS 12127 Study Group. Increasing HIV testing among male partners. AIDS. 2013 Apr 24;27(7):1167-77. doi: 10.1097/QAD.0b013e32835f1d8c. PMID 23343912